CLINICAL TRIAL: NCT00321555
Title: A Phase II Clinical Trial of Anti-Tac(Fv)-PE38 (LMB-2) Immunotoxin for CD25 Positive Hairy Cell Leukemia
Brief Title: LMB-2 to Treat Hairy Cell Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert Kreitman, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060150; 06-C-0150; NCT00337311 (obsolete NCT alias)
Record Dates: First submitted 2006-05-03; First posted 2006-05-04 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Hairy Cell Leukemia
Keywords: Biologic Therapy; Monoclonal Antibody; Immunotherapy; Pseudomonas Exotoxin; Targeted Therapy; Hairy Cell Leukemia; HCL
MeSH Terms: conditions — Leukemia, Hairy Cell | interventions — B3(Fv)-PE38KDEL recombinant immunotoxin; Immunotoxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LMB-2 to Treat Hairy Cell Leukemia (Experimental): LMB-2 Infusion: 40 micro-g/Kg will be infused in 50 ml of 0.9% Sodium chloride (NaCl) and 0.2% albumin via over 30 minutes every other day for 3 doses. Patients may receive up to six treatment cycles every 4 weeks.
  Interventions: Drug: Anti-Tac(Fv)-PE38 (LMB-2) Immunotoxin

INTERVENTIONS:
Drug: Anti-Tac(Fv)-PE38 (LMB-2) Immunotoxin — LMB-2 Infusion: 40 micro-g/Kg will be infused in 50 ml of 0.9% Sodium Chloride (NaCl) and 0.2% albumin via over 30 minutes every other day for 3 doses. Patients may receive up to six treatment cycles every 4 weeks.

SUMMARY:
Background:

* About 80% of patients with hairy cell leukemia (HCL) have tumor cells that have a protein on their surface called cluster of differentiation 25 (CD25).
* The experimental drug LMB-2 is a recombinant immunotoxin that has been shown to kill leukemia and lymphoma cells with the CD25 protein. (A recombinant immunotoxin is a genetically engineered drug that has two parts - a protein that binds or targets a cancer cell, and a toxin that kills the cancer cell to which it binds.)

Objectives:

* To evaluate the safety and effectiveness of LMB-2 in patients with HCL whose cancer cells contain the CD25 protein.
* To evaluate the effects of LMB-2 on the immune system, determine how the drug is metabolized by the body and examine its side effects.

Eligibility:

-Adults with hairy cell leukemia whose tumor cells have CD25 on their surface

Design:

* Up to 27 patients may be included in the study.
* Patients receive an infusion of LMB-2 through a vein every other day for three doses (days 1, 3, 5), constituting one treatment cycle.
* Patients may receive up to six treatment cycles every 4 weeks unless their cancer worsens or they develop unacceptable side effects.
* Blood is drawn weekly for various tests.
* Before each cycle and in follow-up visits, disease status is evaluated with a physical examination, blood tests, chest x-ray and electrocardiogram.
* Before the first cycle, patients may have a computed tomography (CT) scan, echocardiogram (heart ultrasound test) and bone marrow biopsy. With the patient's permission, these tests may be repeated before other cycles also.

DETAILED DESCRIPTION:
Background: About 80% of patients with hairy cell leukemia (HCL) have malignant cells that express cluster of differentiation 25 (CD25) (Tac or Interleukin-2 receptor alpha (IL2Ra)). Normal resting B- and T-cells do not express CD25. LMB-2 is an anti-CD25 recombinant immunotoxin containing variable domains of MAb anti-Tac and truncated Pseudomonas exotoxin. A phase I trial at National Cancer Institute (NCI) found that the maximum tolerated dose (MTD) of LMB-2 was 40 microg/Kg intravenous (IV) given every other day for 3 doses (QOD x3). The most common adverse events were transient fever, hypoalbuminemia and transaminase elevations. In that trial, 4 of 4 patients with chemoresistant HCL had major responses, including one complete (CR) and 3 partial remissions. The patient with CR entered the trial transfusion dependent and now still has normal hemoglobin and platelet counts over 7 years later. Because HCL is more frequently cluster of differentiation 22 (CD22+) than CD25+ (100 vs 80%), HCL patients were subsequently treated with the anti-CD22 recombinant immunotoxin BL22 and no further HCL patients were treated with LMB-2. BL22 has induced 25 CRs out of 51 evaluable HCL patients. LMB-2 may be useful in patients incompletely responding to BL22, because it may distribute more evenly through extravascular sites of disease. Moreover, BL22 but not LMB-2 has caused hemolytic uremic syndrome (HUS) in 7 patients, 6 with HCL, and several of these patients could benefit by LMB-2. Thus, LMB-2 may be a useful and potentially lifesaving agent in patients who are unable to receive or who have not responded adequately to BL22.

Objectives: The purpose of this study is to determine the activity of anti-Tac(Fv)-PE38 (LMB-2) in patients with CD25-expressing hairy cell leukemia (HCL). The primary endpoint of this trial is response rate. We will also evaluate response duration, LMB-2 immunogenicity, pharmacokinetics, toxicity, and monitor soluble Tac levels in the serum.

Eligibility: Patients must have CD25+ HCL cells by flow cytometry, cytopenia or high circulating HCL count, prior treatment with or inability to receive BL22, prior treatment with cladribine, Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2, at least 18 years old, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) grade 0-2, albumin grade 0-1, bilirubin less than or equal to 2.2, creatinine less than or equal to 1.4 or creatinine clearance greater than or equal to 50, lack of high levels of neutralizing antibodies, lack of anti-CD25 Mab therapy for 12 weeks and other systemic treatment for 4 weeks, no prior treatment with LMB-2, lack of other uncontrolled illness including 2nd malignancy, no human immunodeficiency virus (HIV) or hepatitis C positivity, no coumadin therapy, left ventricular ejection fraction (LVEF) greater than or equal to 45%, diffusing capacity of the lungs for carbon monoxide (DLCO) greater than or equal to 55%, and forced expiratory volume 1 (FEV1) greater than or equal to 60%.

Design: Patients will receive LMB-2 at 40 microg/Kg every other day (QOD) x3 at intervals of at least 25 days for up to 6 cycles. Retreatment is permitted in the absence of neutralizing antibodies or progressive disease. Patients in CR may receive 2 consolidation cycles, or 4 consolidation cycles if CR is with minimal residual disease.

Dose level: LMB-2 40 microg/Kg QOD x3

Expected Accrual: 5-10 patients/year, total of 25 patients

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Histopathological evidence of cluster of differentiation 25 (CD25)+ Hairy Cell Leukemia (HCL) confirmed by the National Institutes of Health (NIH) pathology department. This will require a monoclonal population of peripheral malignant lymphocytes that are CD25 positive by fluorescence activated cell sorting (FACS) with anti-CD25 antibody. Positive expression in a FACS assay is defined as more than 2 times the mean fluorescence intensity (MFI) of the control antibody by FACS. HCLv (HCL variant) is usually CD25 negative, and eligibility would require CD25+ HCLv.
  2. At least one of the following indications for treatment: neutropenia (absolute neutrophil count (ANC) less than 1000 cells/ microL), anemia (hemoglobin (Hgb) less than 10g/dL), thrombocytopenia (platelet (Plt) less than 100,000/ microL), an absolute lymphocyte count of greater than 20,000 cells/microL or symptomatic splenomegaly.
  3. Previous treatment with or inability to receive BL22 or HA22 recombinant immunotoxin. Patients must have had at least 2 prior systemic therapies, including 2 courses of a purine nucleoside analog (PNA), or 1 course of either rituximab or BRAF inhibitor following a single prior course of PNA.
  4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.
  5. At least 18 years old.
  6. Understand and give informed consent.
  7. A negative pregnancy test in female patients of childbearing potential. Women must not be breast-feeding.
  8. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 5-times the upper limits of normal. Albumin greater than or equal to 3.0 gm/dL. Total bilirubin less than or equal to 2.2 mg/dL.
  9. Creatinine less than or equal to 1.4 mg/dL or creatinine clearance greater than or equal to 50 ml/min.
  10. Serum that neutralizes less than or equal to 75% of the activity of 1 microg/mL of LMB-2 using a bioassay.
  11. No systemic cytotoxic chemotherapy within 4 weeks of enrollment or systemic steroids (except stable doses of Prednisone less than or equal to 20 mg/day, or up to 4 doses of steroid given for non-therapy reasons) within 4 weeks of enrollment.
  12. No anti-cluster of differentiation 25 (CD25) monoclonal antibody therapy within 12 weeks of enrollment.
  13. No prior treatment with LMB-2.
  14. Patients may not be receiving any other investigational agents.
  15. Patients should not have uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

EXCLUSION CRITERIA:

* Patients who have human immunodeficiency virus (HIV) or hepatitis C. Patients would not be excluded for hepatitis B surface antigen positivity if on Lamivudine.
* Patients receiving coumadin.
* Patients with a left ventricular ejection fraction of less than 45%.
* Patients with a diffusing capacity of the lungs for carbon monoxide (DLCO) less than 55% of normal or an forced expiratory volume 1 (FEV1) less than 60% of normal based on either National Institutes of Health (NIH) or United States of America (USA) normal ranges.
* Patients who have an active 2nd malignancy requiring systemic treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-05-02 (Actual); Primary Completion 2016-08-24 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Kreitman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Background] Carson DA, Wasson DB, Beutler E. Antileukemic and immunosuppressive activity of 2-chloro-2'-deoxyadenosine. Proc Natl Acad Sci U S A. 1984 Apr;81(7):2232-6. doi: 10.1073/pnas.81.7.2232. PMID 6585795
- [Background] Blasinska-Morawiec M, Robak T, Krykowski E, Hellmann A, Urbanska-Rys H. Hairy cell leukemia-variant treated with 2-chlorodeoxyadenosine--a report of three cases. Leuk Lymphoma. 1997 Apr;25(3-4):381-5. doi: 10.3109/10428199709114177. PMID 9168448
- [Background] Cheson BD, Martin A. Clinical trials in hairy cell leukemia. Current status and future directions. Ann Intern Med. 1987 Jun;106(6):871-8. doi: 10.7326/0003-4819-106-6-871. PMID 3555204
- [Derived] Matsushita K, Margulies I, Onda M, Nagata S, Stetler-Stevenson M, Kreitman RJ. Soluble CD22 as a tumor marker for hairy cell leukemia. Blood. 2008 Sep 15;112(6):2272-7. doi: 10.1182/blood-2008-01-131987. Epub 2008 Jul 2. PMID 18596230
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-C-0150.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LMB-2 to Treat Hairy Cell Leukemia
Started | 15
Completed | 9
Not Completed | 6
Not completed — Developed antibodies | 1
Not completed — Switched to alternative treatment | 3
Not completed — Physician Decision | 1
Not completed — Disease progression on study | 1

BASELINE CHARACTERISTICS:
Arm/Group | LMB-2 to Treat Hairy Cell Leukemia
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.49 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Obtain Partial Response/Complete Remission
Description: Partial response requires all of the following for a period of at least 4 weeks: ≥50% decrease in hairy cell count from pretreatment baseline value by flow cytometry. ≥50% reduction in abnormal hepatosplenomegaly by computed tomography or physical exam. No growth in lymphadenopathy. Neutrophils ≥1,500/µL or 50% improvement over baseline without growth factors for at least 4 weeks. Platelets ≥100,000/µL or 50% improvement over baseline. Complete remission requires all of the following: no evidence of leukemic cells by routine hematoxylin and eosin stains of the peripheral blood and bone marrow. No hepatomegaly, splenomegaly, or lymphadenopathy (not >2 cm in short axis) by physical examination and appropriate radiographic techniques. Normal complete blood count as exhibited by Neutrophils ≥1,500/µL, Platelets ≥100,000/µL, and Hemoglobin ≥11.0g/dL without transfusions or growth factors for at least 4 weeks.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | LMB-2 to Treat Hairy Cell Leukemia
Number analyzed (Participants) | 15
Participants
  Complete Remission | 1
  Partial Response | 5

2. Secondary Outcome: Duration of Response
Description: Duration of response is the duration that the patients qualifies for at least a Partial Response (PR). Partial response requires all of the following for a period of at least 4 weeks: ≥50% decrease in hairy cell count from pretreatment baseline value by flow cytometry. ≥50% reduction in abnormal hepatosplenomegaly by computed tomography or physical exam. No growth in lymphadenopathy. Neutrophils ≥1,500/µL or 50% improvement over baseline without growth factors for at least 4 weeks. Platelets ≥100,000/µL or 50% improvement over baseline. Hemoglobin ≥11.0 g/dL or 50% improvement over baseline without transfusions or growth factors for at least 4 weeks.
Time Frame: Participants were assessed at 5.0658, 12.0066, 20.1645, 26.9079, 35.0987, and 45.1316 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LMB-2 to Treat Hairy Cell Leukemia
Number analyzed (Participants) | 6
months | 23.5 [5.1 to 45.1]

3. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 83 months and 15 days.
Measure: Count of Participants; unit: Participants
Arm/Group | LMB-2 to Treat Hairy Cell Leukemia
Number analyzed (Participants) | 15
Participants | 13

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 83 months and 15 days.
Arm/Group | LMB-2 to Treat Hairy Cell Leukemia
All-Cause Mortality (participants affected / at risk) | 2/15
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMB-2 to Treat Hairy Cell Leukemia (N=15)
Allergic reaction (Immune system disorders) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1)
Death NOS (General disorders) | 2 (2)
Vasovagal reaction (Nervous system disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMB-2 to Treat Hairy Cell Leukemia (N=15)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (9)
Allergic reaction (Immune system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 5 (12)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (11)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 1 (2)
Chills (General disorders) | 1 (2)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine increased (Investigations) | 1 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema face (General disorders) | 2 (4)
Edema limbs (General disorders) | 7 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 3 (6)
Haptoglobin decreased (Investigations) | 2 (2)
Headache (Nervous system disorders) | 4 (4)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (3)
Hypertension (Vascular disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (26)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (5)
Hyponatremia (Metabolism and nutrition disorders) | 5 (9)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2)
Investigations - Other, Bicarbonate serum low (Investigations) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (10)
Neutrophil count decreased (Investigations) | 3 (4)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 4 (10)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vascular disorders - Other, Vascular leak syndrome (Vascular disorders) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight gain (Investigations) | 4 (5)
White blood cell decreased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT00321555/Prot_SAP_004.pdf
  • Informed Consent Form (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT00321555/ICF_003.pdf